CLINICAL TRIAL: NCT05135884
Title: Lucerne Fall Risk Prediction Score for Stroke Rehabilitation
Acronym: L-PRESTO
Status: Completed | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Janne Veerbeek, Principal Investigator, Luzerner Kantonsspital
Other Study IDs: L-PRESTO
Record Dates: First submitted 2021-11-04; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort
  Interventions: Behavioral: Standard inpatient stroke rehabilitation

INTERVENTIONS:
Behavioral: Standard inpatient stroke rehabilitation — According to Swiss national guidelines and local protocols

SUMMARY:
In Switzerland, every year around 16'000 people suffer a stroke. Stroke represents the third most common cause of death in Switzerland and leads to impairments (e.g., motoric, cognitive, sensory) resulting in disability. People with disabilities after stroke should have access to specialised interprofessional rehabilitation settings.

During inpatient rehabilitation, 15-36% of the patients experience one or more falls. It is well known that stroke is an important risk factor for falls. On average stroke patients fall 1.77 times more than the age- and gender-matched controls over 13 months. Falling events during inpatient stroke rehabilitation result in an extension of rehabilitation stay of about eleven days. Wong et al. (2016) suspect that a reduction in the activity level due to falls, fear of falling again as well as changes in discharge conditions could be the reason for this extended length of stay. Walsh et al. (2018) demonstrate that patients who fall once within the first year after stroke cause € 8'600 and recurrent fallers € 12'700 higher healthcare costs.

Fall risk factors after stroke are well investigated. Campbell & Matthews (2010) have collected multiple factors for falls in inpatient stroke rehabilitation from 1990 to 2009 in an integrative review. A newer systematic review points out physical function, hemi-attention, and stability as the most important factors for falls in inpatient stroke rehabilitation. However, none of the included studies showed a validated prediction model with acceptable performance. Hence, further investigations regarding the impact of various valid and reliable fall risk assessments at admission in inpatient rehabilitation are needed.

The neurorehabilitation team of LUKS systematically assesses the patient's functions and activity to design patient-specific, evidence-based rehabilitation. Therefore, a population-specific fall risk model based on standardized assessments performed in the clinical routine would help to identify patients with a high risk of falling during rehabilitation without the need of implementing an existing model with a low performance.

Aim of the study The main aim of this study is to establish a multivariable prediction model for falls during inpatient rehabilitation in acute and subacute stroke patients admitted to the Clinic for Neurology and Neurorehabilitation of the Kantonsspital Luzern (LUKS) in Lucerne, Switzerland.

The secondary aim is to explore the value of the mini-BESTest as a fall predictor in a subgroup consisting of patients who are ambulatory at admission to the Clinic for Neurology and Neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Acute/ subcute first or recurrent stroke
* Inpatient rehabilitation
* Signed general consent

Exclusion Criteria:

- Re-rehabilitation due to a chronic stroke

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patiets admitted to inpatient neurorehabilitation after an acute stroke
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Occurance of at least one fall | During inpatient stroke rehabilitation, an average of 6 weeks
  Event of least one fall (yes/ no) during inpatient stroke rehabilitation

SECONDARY OUTCOMES:
Lucerne ICF Based Multidisciplinary Observational Scale (45-225 points, higher scores being better) | Rehabilitation admission
  Activities of daily living
Functional Independence Measure (18-126 points, higher scores being better) | Rehabilitation admission
  Activities of daily living
Montreal Cognitive Assessment (0-30 points, higher scores being better) | Rehabilitation admission
  Cognitive function
Apraxia Screen of Tulia (0-12 points, higher scores being better) | Rehabilitation admission
  Apraxia
Mini Balance Evaluation Systems Test (0-28 points, higher scores being better) | Rehabilitation admission
  Balance
2-Minute Walk Test (meter, higher scores being better) | Rehabilitation admission
  Gait speed and walking distance
Timed up and go (seconds, lower scores being better) | Rehabilitation admission
  Mobility
Catherine Bergego Scale (0-30 points, lower scores being better) | Rehabilitation admission
  Visuospatial function
Language Screening Test (0-15 points, higher scores being better) | Rehabilitation admission
  Speech function

CONTACTS AND LOCATIONS:
Overall Officials: Janne M. Veerbeek, PhD, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Breisinger TP, Skidmore ER, Niyonkuru C, Terhorst L, Campbell GB. The Stroke Assessment of Fall Risk (SAFR): predictive validity in inpatient stroke rehabilitation. Clin Rehabil. 2014 Dec;28(12):1218-24. doi: 10.1177/0269215514534276. Epub 2014 May 21. PMID 24849795
- [Background] Campbell GB, Matthews JT. An integrative review of factors associated with falls during post-stroke rehabilitation. J Nurs Scholarsh. 2010 Dec;42(4):395-404. doi: 10.1111/j.1547-5069.2010.01369.x. Epub 2010 Oct 13. PMID 21091622
- [Background] Flamand-Roze C, Falissard B, Roze E, Maintigneux L, Beziz J, Chacon A, Join-Lambert C, Adams D, Denier C. Validation of a new language screening tool for patients with acute stroke: the Language Screening Test (LAST). Stroke. 2011 May;42(5):1224-9. doi: 10.1161/STROKEAHA.110.609503. Epub 2011 Apr 12. PMID 21487118
- [Background] Meyer K, Simmet A, Arnold M, Mattle H, Nedeltchev K. Stroke events, and case fatalities in Switzerland based on hospital statistics and cause of death statistics. Swiss Med Wkly. 2009 Feb 7;139(5-6):65-9. doi: 10.4414/smw.2009.12448. PMID 19204838
- [Background] National Institute for Health and Care Excellence. Stroke rehabilitation in adults. 2013. https://www.nice.org.uk/guidance/cg162/chapter/1-Recommendations#organising-health-and-social-care-for-people-needing-rehabilitation-after-stroke
- [Background] Nyberg L, Gustafson Y. Patient falls in stroke rehabilitation. A challenge to rehabilitation strategies. Stroke. 1995 May;26(5):838-42. doi: 10.1161/01.str.26.5.838. PMID 7740577
- [Background] Persson CU, Kjellberg S, Lernfelt B, Westerlind E, Cruce M, Hansson PO. Risk of falling in a stroke unit after acute stroke: The Fall Study of Gothenburg (FallsGOT). Clin Rehabil. 2018 Mar;32(3):398-409. doi: 10.1177/0269215517728325. Epub 2017 Sep 11. PMID 28891685
- [Background] Simpson LA, Miller WC, Eng JJ. Effect of stroke on fall rate, location and predictors: a prospective comparison of older adults with and without stroke. PLoS One. 2011 Apr 29;6(4):e19431. doi: 10.1371/journal.pone.0019431. PMID 21559367
- [Background] Walsh ME, Horgan NF, Walsh CD, Galvin R. Systematic review of risk prediction models for falls after stroke. J Epidemiol Community Health. 2016 May;70(5):513-9. doi: 10.1136/jech-2015-206475. Epub 2016 Jan 14. PMID 26767405
- [Background] Walsh ME, Sorensen J, Galvin R, Williams DJ, Harbison JA, Murphy S, Collins R, McCabe DJ, Crowe M, Horgan NF. First year post-stroke healthcare costs and fall-status among those discharged to the community. Eur Stroke J. 2018 Sep;3(3):254-262. doi: 10.1177/2396987318764954. Epub 2018 Mar 15. PMID 31008356
- [Background] Wong JS, Brooks D, Mansfield A. Do Falls Experienced During Inpatient Stroke Rehabilitation Affect Length of Stay, Functional Status, and Discharge Destination? Arch Phys Med Rehabil. 2016 Apr;97(4):561-566. doi: 10.1016/j.apmr.2015.12.005. Epub 2015 Dec 19. PMID 26711169